CLINICAL TRIAL: NCT02311608
Title: Comparative Effectiveness Research: Effects of Terlipressin When Usual Somatostatin or Octreotide Dose Fails to Treat the Patients With Acute Variceal Bleeding
Brief Title: Effects of Terlipressin When Usual Somatostatin or Octreotide Dose Fails
Acronym: CER:T
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department fo Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Other Study IDs: CSY-LB2-2014
Record Dates: First submitted 2014-11-26; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices; Hemorrhage
Keywords: acute variceal hemorrhage; terlipressin; somatostatin; octreotide; comparative effectiveness research
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices; Hemorrhage | interventions — Terlipressin; Octreotide; Somatostatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- High Dose Somatostatin/Octreotide: continuous IV infusion of 500μg/h of Somatostatin or continuous IV infusion of 50μg/h of Octreotide when usual somatostatin or Octreotide dose fails to achieve hemostasis of acute variceal bleeding patients
  Interventions: Drug: Usual Dose Somatostatin/Octreotide; Drug: High Dose Somatostatin/Octreotide
- Terlipressin as salvage: an initial injection of 2mg of Terlipressin followed by an injection of 1mg of Terlipressin per 6h when usual somatostatin or Octreotide dose fails to achieve hemostasis of acute variceal bleeding patients
  Interventions: Drug: Terlipressin; Drug: Usual Dose Somatostatin/Octreotide
- Terlipr+usual dose somato/Octreo: an initial injection of 2mg of Terlipressin followed by an injection of 1mg of Terlipressin per 6h together with continuous IV infusion of 250μg/h of Somatostatin or continuous IV infusion of 25μg/h of Octreotide when usual somatostatin or Octreotide dose fails to achieve hemostasis of acute variceal bleeding patients
  Interventions: Drug: Terlipressin; Drug: Usual Dose Somatostatin/Octreotide; Drug: High Dose Somatostatin/Octreotide
- Control:Usual Dose Somato/Octreo: Hemostasis achieved by continuous IV infusion of 250μg/h of Somatostatin or continuous IV infusion of 25μg/h of Octreotide
  Interventions: Drug: Usual Dose Somatostatin/Octreotide
- Control: Initial Terlipressin: Hemostasis achieved by an initial injection of 2mg of Terlipressin followed by an injection of 1mg of Terlipressin per 6h
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — administered as a first-line medicine or as salvage
  Other Names: Hanwei
  Groups: Control: Initial Terlipressin; Terlipr+usual dose somato/Octreo; Terlipressin as salvage
Drug: Usual Dose Somatostatin/Octreotide — administered as a first-line medicine or as salvage
  Other Names: Yisuo/Shanning
  Groups: Control:Usual Dose Somato/Octreo; High Dose Somatostatin/Octreotide; Terlipr+usual dose somato/Octreo; Terlipressin as salvage
Drug: High Dose Somatostatin/Octreotide — administered as salvage
  Other Names: Yisuo/Shanning
  Groups: High Dose Somatostatin/Octreotide; Terlipr+usual dose somato/Octreo

SUMMARY:
To observe and access the Effects and safety of terlipressin or high dose somatostatin/octreotide when usual dose somatostatin/octreotide fail to achieve hemostasis in patients with acute variceal bleeding.

DETAILED DESCRIPTION:
The prognosis information of the patients with acute variceal bleeding will be collected, including hemostasis rate, early rebleeding rate, mortality, complications, severity adverse events, economic burdens and quality of life, when terlipressin or high dose somatostatin/octreotide is used as salvation to patients fail to achieve initial hemostasis.The results may help gastroenterologists to make decisions when administering vasoactive medicines to those suffered from acute variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis patients admitted to Emergency Department because of acute variceal bleeding

Exclusion Criteria:

* No signs of variceal bleeding are found by endoscopy or portal hypertensive gastropathy is responsible for the bleeding
* Patients undergo endoscopy after 72h from the beginning of acute variceal bleeding
* Patients with hepatorenal syndrome
* Patients with ischemia organic cardiopathy (including myocardial infarction or unstable angina pectoris) or myocardial ischemia indicated by ECG in the past 6 months
* Patients allergic to/with contraindications of vasoactive drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cirrohsis patients with acute variceal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The Change of Rebleeding Rate | 1month, 3months, 6 months, 12 months

SECONDARY OUTCOMES:
Economic Cost | up to 12 months
The Change of Quality of Life | 1month, 3months, 6 months, 12 months
The Change of Survival Rate | 1month, 3months, 6 months, 12 months
The Change of Complication Rate | 1month, 3months, 6 months, 12 months
The Change of Drug Adverse Reaction Rate | 1month, 3months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Azam Z, Hamid S, Jafri W, Salih M, Abbas Z, Abid S, Shah H. Short course adjuvant terlipressin in acute variceal bleeding: a randomized double blind dummy controlled trial. J Hepatol. 2012 Apr;56(4):819-24. doi: 10.1016/j.jhep.2011.11.019. Epub 2011 Dec 16. PMID 22178268
- [Background] Kalambokis G, Economou M, Paraskevi K, Konstantinos P, Pappas C, Katsaraki A, Tsianos EV. Effects of somatostatin, terlipressin and somatostatin plus terlipressin on portal and systemic hemodynamics and renal sodium excretion in patients with cirrhosis. J Gastroenterol Hepatol. 2005 Jul;20(7):1075-81. doi: 10.1111/j.1440-1746.2005.03902.x. PMID 15955217
- [Background] Romero G, Kravetz D, Argonz J, Bildozola M, Suarez A, Terg R. Terlipressin is more effective in decreasing variceal pressure than portal pressure in cirrhotic patients. J Hepatol. 2000 Mar;32(3):419-25. doi: 10.1016/s0168-8278(00)80392-x. PMID 10735611
- [Background] Lo GH, Perng DS, Chang CY, Tai CM, Wang HM, Lin HC. Controlled trial of ligation plus vasoconstrictor versus proton pump inhibitor in the control of acute esophageal variceal bleeding. J Gastroenterol Hepatol. 2013 Apr;28(4):684-9. doi: 10.1111/jgh.12107. PMID 23278466
- [Background] Sola E, Lens S, Guevara M, Martin-Llahi M, Fagundes C, Pereira G, Pavesi M, Fernandez J, Gonzalez-Abraldes J, Escorsell A, Mas A, Bosch J, Arroyo V, Gines P. Hyponatremia in patients treated with terlipressin for severe gastrointestinal bleeding due to portal hypertension. Hepatology. 2010 Nov;52(5):1783-90. doi: 10.1002/hep.23893. PMID 20931555
- [Background] Abid S, Jafri W, Hamid S, Salih M, Azam Z, Mumtaz K, Shah HA, Abbas Z. Terlipressin vs. octreotide in bleeding esophageal varices as an adjuvant therapy with endoscopic band ligation: a randomized double-blind placebo-controlled trial. Am J Gastroenterol. 2009 Mar;104(3):617-23. doi: 10.1038/ajg.2008.147. Epub 2009 Feb 17. PMID 19223890
- [Background] Lo GH, Chen WC, Wang HM, Lin CK, Chan HH, Tsai WL, Cheng LC, Yu HC, Tsay FW. Low-dose terlipressin plus banding ligation versus low-dose terlipressin alone in the prevention of very early rebleeding of oesophageal varices. Gut. 2009 Sep;58(9):1275-80. doi: 10.1136/gut.2008.165910. Epub 2009 Apr 21. PMID 19386609
- [Background] Fabrizi F, Dixit V, Martin P. Meta-analysis: terlipressin therapy for the hepatorenal syndrome. Aliment Pharmacol Ther. 2006 Sep 15;24(6):935-44. doi: 10.1111/j.1365-2036.2006.03086.x. PMID 16948805
- [Background] D'Amico G, Pietrosi G, Tarantino I, Pagliaro L. Emergency sclerotherapy versus vasoactive drugs for variceal bleeding in cirrhosis: a Cochrane meta-analysis. Gastroenterology. 2003 May;124(5):1277-91. doi: 10.1016/s0016-5085(03)00269-5. PMID 12730868
- [Background] Escorsell A, Ruiz del Arbol L, Planas R, Albillos A, Banares R, Cales P, Pateron D, Bernard B, Vinel JP, Bosch J. Multicenter randomized controlled trial of terlipressin versus sclerotherapy in the treatment of acute variceal bleeding: the TEST study. Hepatology. 2000 Sep;32(3):471-6. doi: 10.1053/jhep.2000.16601. PMID 10960437
- [Result] Baik SK, Jeong PH, Ji SW, Yoo BS, Kim HS, Lee DK, Kwon SO, Kim YJ, Park JW, Chang SJ, Lee SS. Acute hemodynamic effects of octreotide and terlipressin in patients with cirrhosis: a randomized comparison. Am J Gastroenterol. 2005 Mar;100(3):631-5. doi: 10.1111/j.1572-0241.2005.41381.x. PMID 15743362
- [Result] Villanueva C, Planella M, Aracil C, Lopez-Balaguer JM, Gonzalez B, Minana J, Balanzo J. Hemodynamic effects of terlipressin and high somatostatin dose during acute variceal bleeding in nonresponders to the usual somatostatin dose. Am J Gastroenterol. 2005 Mar;100(3):624-30. doi: 10.1111/j.1572-0241.2004.40665.x. PMID 15743361